CLINICAL TRIAL: NCT00211783
Title: fMRI for the Study of Response Inhibition, and Face and Linguistic Processing in Autism
Brief Title: Functional Magnetic Resonance Imaging (fMRI) for the Study of Response Inhibition, and Face and Linguistic Processing in Autism
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO# 04-0749
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Autism; Asperger's Syndrome
Keywords: autism; fMRI; response inhibition; face processing; linguistic processing
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Autism
  Interventions: Procedure: fMRI
- Control

INTERVENTIONS:
Procedure: fMRI — there is no intervention
  Groups: Autism

SUMMARY:
This study investigates face processing, response inhibition and phoneme processing in autistic adults by fMRI.

DETAILED DESCRIPTION:
Fifteen adult outpatients with high functioning autism or Asperger's Syndrome will be recruited. Fifteen healthy volunteers matched for age and IQ will also be recruited. Participants will undergo an fMRI scan. During the scan they will perform a task. The paradigm is designed to test control inhibition, face processing and language. Therefore, it includes a go-no go test, a face emotion discrimination test and a linguistic sound. The subjects are shown a series of faces with happy or sad expressions in random order. Each face presentation is accompanied by either a standard or variant sound. The sound stimulus is the English phoneme /oe/. The variant sound was created by raising the frequency of the standard sound by 20%. The task consists of four blocks. During each block the subjects are asked to press a button when they see a happy or sad face depending on the block. Each block consists of 96 trials lasting 2 seconds and an initial and final fixation period of 40 sec. For each trial the target image is projected for 500 ms. There is 1250 ms fixation time allowed for response and 250 ms for jitter. Twenty-four of the 96 trials are no go trials and 16/96 are sound oddball trials. The oddball is at least two trials apart (between two variant sounds there are at least two standard sounds). There are 24 faces displayed in total, 12 female and 12 male. Faces switch every 16 trials. Face genders are balanced. The faces were selected with over 80% congruency except for two faces with congruency of over 72%. The correlation between sound (2 conditions: standard versus variant) and target condition (go-no go) is zero. The task was piloted on healthy controls and autistic adults. All subjects performed well.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 18-50 years old
* Diagnosis: autism spectrum disorder by Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) and Autism Diagnostic Interview - Revised (ADI-R)
* Intelligence quotient (IQ) > 80
* Outpatients

Exclusion Criteria:

* Subjects with epilepsy
* Subjects with history of schizophrenia, schizoaffective disorder or other Axis 1 mental disorders, such as bipolar disorder
* Subjects reporting history of encephalitis, phenylketonuria, tuberous sclerosis, fragile X syndrome, anoxia during birth, neurofibromatosis, hypomelanosis of Ito, hypothyroidism, Duchenne muscular dystrophy, and maternal rubella
* Subjects who have received depot neuroleptic medication, or other psychoactive drugs within the past 5 weeks.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Thirty adults with ASD and 30
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2004-11; Primary Completion 2011-11 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
BOLD | at single study visit
  Differences in BOLD betweens controls and ASD group BOLD - blood-oxygen-level-dependent contrast

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Anagnostou, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States